

### INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

TITLE: Phase I/II Study of Oral ONC201 in Patients with Relapsed

or Refractory Acute Leukemias and High-Risk

Myelodysplastic Syndromes

**PROTOCOL NO.:** 2014-0731

WCG IRB Protocol #20152152

**SPONSOR:** The University of Texas MD Anderson Cancer Center

**INVESTIGATOR:** Gautam Borthakur, MBBS

1515 Holcombe Blvd., Unit 428

Houston, Texas 77030

**United States** 

STUDY-RELATED

PHONE NUMBER(S): Gautam Borthakur, MBBS

713-563-1586

713-792-2121 (24-hours)

Participant's Name Medical Record Number

Tartiopant's Name Wedical Record Number

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

### STUDY SUMMARY

You are being asked to take part in this study because you have acute myelogenous leukemia (AML), acute lymphoblastic leukemia (ALL), or high-risk myelodysplastic syndrome (MDS) that is relapsed (has come back), is refractory (has not responded to treatment) or have untreated high risk MDS or acute leukemia but are not eligible for more intensive therapies (Phase I Arm E and Phase II only).

There are 2 parts to this clinical research study: Phase I (Dose Escalation) and Phase II (Dose Expansion).

The goal of Phase I of this clinical research study is to find the highest tolerable dose of ONC201 that can be given alone or in combination with venetoclax to patients with relapsed or refractory AML, ALL, or MDS.

The goal of Phase II of this study is to learn if the dose of ONC201 that is found in Phase I given alone or in combination with venetoclax can help to control the disease.

The safety of ONC201 given alone or in combination with venetoclax will be studied in both phases of this study.

This is the first study using ONC201 in humans.

ONC201 is in a very early stage of development for use in humans. Providing direct medical benefit to you is not the purpose of this study. While Phase II will look at the effectiveness of the study drug, the main purpose of this study is to learn about the safety of the drug. Please carefully read the sections on risk and benefits below.

This is an investigational study. ONC201 is not FDA approved or commercially available. It is currently being used for research purposes only. Venetoclax is FDA approved and commercially available for the treatment of AML and chronic lymphocytic leukemia/small lymphocytic lymphoma. It is considered investigational to give ONC201 and venetoclax together. The study doctor can explain how the study drugs are designed to work.

Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment. You may not want to take part in this study because it is the first study of ONC201 in humans.

You can read a full list of potential side effects below in the Possible Risks section of this consent.

You may continue taking the study drug(s) for as long as the doctor thinks it is in your best interest.

ONC201 will be provided at no cost to you while you are on study. You and/or your insurance provider will be responsible for the cost of venetoclax, if you receive it.

You may choose not to take part in this study. You may choose to receive chemotherapy and/or other FDA-approved drugs. Depending on what kind of cancer you have, you could receive azacitidine or decitabine. You may choose to receive other investigational therapies, if available. You may choose not to have treatment for cancer at all. If you decide that you don't want any more active treatment, one of your options is called "comfort care." Comfort care includes pain medication and other support. It aims

to maintain your comfort and dignity rather than cure disease. Usually, this care can be provided at home.

If you think you might prefer comfort care, please discuss this with your family, friends, and your doctor.

In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

### 1. STUDY DETAILS

## **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. The following screening tests will be performed within 28, 14, and 7 days before your first dose of study drug, to help the doctor decide if you are eligible:

# Within **28 days** before your first dose:

- Your medical history and your height will be collected.
- You will have an electrocardiogram (EKG) to check your heart function.
- You will have a bone marrow aspirate or biopsy for cytogenetic testing. To collect a bone marrow aspirate/biopsy, an area of the hip or other site is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. Cytogenetic testing looks at how genetic changes to cells may affect how the disease may react to the study drug.

### Within **14 days** before your first dose:

- Your ECOG status and weight will be collected.
- Blood (about 2 tablespoons) and urine will be collected for routine tests.
- You will have a chest x-ray to check the condition of your lungs.
- You will have a neurological exam (tests to check the functioning of your nerves, including tests of your balance and reflexes). If you have neurological symptoms at any other point in this study, this exam may be repeated.
- If you did not have one at your first screening visit, you will have a bone marrow aspirate/biopsy for pharmacodynamic (PD) and cytogenetic testing. PD testing measures how the level of study drug in your body may affect the disease.
- You will have a bone marrow aspirate to check for any genetic mutations (a type of genetic change). If the doctor thinks it is needed, you may have blood (about 1 teaspoon) drawn for this testing instead.

### Within **7 days** before your first dose:

- You will have a physical exam, including vital signs and medical history review.
- Blood (about 2-3 tablespoons) will be collected for routine tests. This routine blood draw will include a pregnancy test if you can become pregnant. To take part in this study, you cannot be pregnant.
- Blood (about 2 teaspoons) will be drawn for pharmacokinetic (PK) and PD testing. PK testing measures the amount of study drug in the body. This sample

is drawn so researchers can compare the results to future PK testing in this study.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.

### **Study Groups**

If you are found to be eligible to take part in this study, you will be enrolled in a study group (Arm) based on the type of disease you have and/or when you joined this study. Up to 120 participants will be enrolled in Phase I of the study, and up to 36 participants will be enrolled in Phase II. All will take part at MD Anderson.

If you are enrolled in **Phase I Arms A, B, C, D, E, or F,** the dose and frequency of ONC201 you receive will depend on when you join the study. The first group of participants will receive the lowest dose level of ONC201. If no intolerable side effects are seen, the next group of participants will receive a higher dose than the group before them. This will continue until the highest tolerable dose of ONC201 is found. The dose you receive may be too low to have an effect on your disease, or so high that it causes bad side effects.

If you are enrolled in **Phase I Arm F**, you will also receive venetoclax. It is planned for all participants in Arm F to receive the same standard dose of venetoclax.

If you are enrolled in **Phase II**, you will receive ONC201 at the highest dose level that was tolerated by participants in the Phase I portion of the study.

### **Study Drug Administration**

In Arms A, B, C, D and E, each study drug cycle is 21 days. If you are enrolled in Phase I Arm F or Phase II, each cycle will be 28 days.

You will take ONC201 capsules by mouth as directed by your doctor 2 hours before or 1 hour after a meal. If you vomit after taking ONC201, you should not retake the dose. Your doctor will tell you how many capsules to take and how often to take them (either 1 or 2 times every week, depending on what group you are assigned to). You should take each dose at about the same time of day, each day you are assigned to take it. You must not crush or chew the capsules or dissolve them in liquid.

You will be given a study drug diary to write down any missed doses. You will give your study drug diary to the study doctor at each clinic visit.

Your dose may be increased or decreased if you have any side effects, if you respond to the study drug, or if the doctor thinks that the next higher dose level is safe.

If you are in Arm F, you will also take venetoclax every day on Days 1-21 of each 28-day cycle.

You will no longer be able to take the study drug(s) if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the end-of-study visit.

## **Study Visits – All Participants**

All participants will have the following tests and procedures:

## On Day 1 of Cycle 1:

- You will have a physical exam, including vital signs, weight, and discussion about any other medications you are taking.
- You will receive additional instructions about neurological side effects and precautions you should take during this study.
- Blood (about 2 tablespoons) will be drawn for routine tests.
- You will have 1 EKG before your dose of ONC201 and then 3 more times over the next 2 hours after the first dose.

On Days 2 Cycle 1, you will have an EKG.

### On Days 8 and 15 of Cycle 1:

- Blood (about 2 tablespoons) will be drawn for routine tests.
- You will have an EKG, vital signs, and discussion about any other medications you are taking.

## On Day 22 of Cycle 1 (Arm E only):

Blood (about 2 tablespoons) will be drawn for routine tests.

### On **Day 1 of Cycles 2 and beyond**:

- You will have a physical exam, including vital signs and a discussion of any other medications you are taking.
- You will have an EKG before your dose of study drug.
- Blood (about 2 tablespoons) will be drawn for routine tests.
- Blood (about 2 teaspoons) will be drawn for PD testing.
- On Cycle 2 only, you will have a bone marrow aspirate/biopsy for PD testing.

On **Day 21 of Cycle 3, and then any time the doctor thinks it is needed after that**, you will have a bone marrow aspirate/biopsy for cytogenetic, biomarker, and PD testing. Biomarkers are found in the blood/tissue and may be related to your reaction to the study drug.

# Study Visits - Phase I Arm A Only

In addition to the tests and procedures described in the "Study Visits - All Participants" section above, participants in Phase I Arm A will also have the following:

**During Cycle 1 only**, blood (about 1 teaspoon each time) will be drawn for PD testing before your first dose of ONC201 and then at about 24 hours, 72 hours, and 7 days after the first dose.

**During Cycle 1 only**, blood (about 1 teaspoon each time) will be drawn for PK testing:

- Before your first dose of ONC201 and then 4 more times over the 6 hours after the dose;
- At about 24 hours, 2 days, 4 days, and 7 days after your first dose of ONC201;
   and
- Before your second dose of ONC201.

## Study Visits - Phase I Arm B Only

In addition to the tests and procedures described in the "Study Visits - All Participants" section above, participants in Phase I Arm B will also have the following:

**During Cycle 1 only**, blood (about 1 teaspoon each time) will be drawn for PD testing before your first dose of ONC201 and then at about 24 hours, 72 hours, and 7 days after the first dose.

**During Cycles 1 and 2 only**, blood (about 1 teaspoon each time) will be drawn for PK testing:

- Before your first dose of ONC201 and then 4 more times over the 6 hours after the dose;
- At about 24 hours, 2 days, and 4 days after your first dose of ONC201; and
- Before your second dose of ONC201.

### Study Visits – Phase I Arms C and E Only

In addition to the tests and procedures described in the "Study Visits - All Participants" section above, participants in Phase I Arms C and E will also have the following:

**During Cycle 1 only**, blood (about 1 teaspoon each time) will be drawn for PD testing before your first dose of ONC201 and then at about 24 hours, 72 hours, and 7 days after the first dose.

**During Cycles 1 and 2 only**, blood (about 1 teaspoon each time) will be drawn for PK testing:

- Before your first and second dose of ONC201 and then 4 more times over the 6 hours after the dose; and
- At about 24 hours, 2 days, and 3 days after your first and second dose of ONC201,

## Study Visits - Phase I Arm D Only

In addition to the tests and procedures described in the "Study Visits - All Participants" section above, participants in Phase I Arm D will also have the following:

**During Cycle 1 only**, blood (about 1 teaspoon each time) will be drawn for PD testing before your first dose of ONC201 and then at about 24 hours, 72 hours, and 7 days after the first dose.

**During Cycles 1 and 2 only**, blood (about 1 teaspoon each time) will be drawn for PK testing:

- Before your first dose of ONC201 on Days 1 and 2 and then 4 more times over the 6 hours after the dose; and
- Before the second dose of ONC201 on Day 1 and then 2 more times over the 2 hours after the dose.

# Study Visits - Phase I Arm F Only

In addition to the tests and procedures described in the "Study Visits - All Participants" section above, participants in Phase I Arm F will also have the following:

**During Cycle 1 only**, blood (about 1 teaspoon each time) will be drawn for PD testing:

- Before your first dose of venetoclax on Day 1;
- On Day 4, at about 72 hours after the first dose of venetoclax and before you take your dose of ONC201;
- On Day 7; and
- On Days 11 and 18 before taking the study drugs.

**During Cycle 1 only**, blood (about 1 teaspoon each time) will be drawn for PK testing:

- Before your dose of ONC201 on Days 4 and 5 and then 4 more times over the 6 hours after the dose;
- At about 24 hours, 2 days, and 4 days after the second dose; and
- On Day 11.

**During Cycle 2 only**, blood (about 1 teaspoon each time) will be drawn for PK testing:

- Before your dose of ONC201 on Days 3 and 4 and then 4 more times over the 6 hours after the dose:
- At about 24 hours, 2 days, and 4 days after the second dose; and
- On Day 11.

# **End-of-Study Visit**

About 1 month after your last dose of study drug:

- You will have a physical exam, including vital signs and a discussion of any other medications you are taking.
- You will have an EKG.
- Blood (about 2 tablespoons) will be drawn for routine tests.

- If the doctor thinks it is needed, blood (about 2 teaspoons) will be drawn for PK and PD testing.
- If the doctor thinks it is needed, you will have a bone marrow aspirate/biopsy to check for any genetic mutations.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. These side effects will vary from person to person. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You should discuss these with the study doctor. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death.

Tell the study staff about any side effects you may have, even if you do not think they are related to the study drug/procedures.

ONC201 and venetoclax each may cause low blood cell counts (red blood cells, platelets, and/or white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become lifethreatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

## **ONC201 Side Effects**

This is an early study of ONC201 in humans, so the side effects are not well known. Based on results of early studies in humans, ONC201 may cause:

- fatigue
- decreased brain function (possible paralysis and/or coma)
- seizure
- stroke
- headache
- difficulty waking
- difficulty forming or speaking words
- difficulty sleeping
- weakness on one side

- nausea
- vomiting
- diarrhea
- intestinal blockage
- low blood levels of phosphate (possible bone damage)
- high blood sugar (possible diabetes)
- low blood cell count (red/white)
- bleeding

- muscle weakness
- difficulty breathing
- breakdown products of the cancer cells entering the blood stream (possible weakness, low blood pressure, muscle cramps, kidney damage, and/or other organ damage)
- severe life-threatening

## Venetoclax Side Effects

# Common (occurring in more than 20% of patients)

| <ul> <li>swelling (arm/leg)</li> <li>fatigue</li> <li>high blood sugar (possible diabetes)</li> <li>abnormal salts, minerals, and/or acids in the blood (possible weakness, swelling, fatigue, low blood pressure, organ failure, heart problems, changes in mental status, and/or seizure)</li> </ul> | <ul> <li>diarrhea</li> <li>nausea</li> <li>low blood counts (red, platelets, and white)</li> <li>abnormal liver tests (possible liver damage)</li> </ul> | <ul> <li>muscle and/or bone pain</li> <li>upper respiratory tract infection</li> <li>cough</li> </ul> |
|---|---|---|
|---|---|---|

# Occasional (occurring in 3-20% of patients)

| fever | <ul> <li>abdominal pain</li> </ul> | <ul> <li>difficulty breathing</li> </ul> |
|---|---|---|
| <ul><li>headache</li></ul> | <ul> <li>mouth blisters/sores</li> </ul> | <ul> <li>severe life-threatening</li> </ul> |
| <ul><li>dizziness</li></ul> | (possible difficulty | infection (possible low |
| skin rash | swallowing) | blood pressure, kidney |
| vomiting | joint pain | failure, and/or heart |
| constipation | <ul> <li>pneumonia</li> </ul> | failure) |

## Rare but serious (occurring in fewer than 3% of patients)

• tumor lysis syndrome (TLS)

TLS is a problem that can occur when cancer cells break down rapidly and the body has to get rid of the broken up cell parts. Sometimes your body, especially the kidneys, cannot remove the cell parts quickly enough, so the level of some of these cell products in your blood, such as salts and acids, can rise. This can happen especially in participants with large tumors or a high number of cancerous white cells in the blood. TLS can lead to serious problems, such as effects on your kidneys and heart (including abnormal heart rhythms), seizures, or even death.

If you develop TLS, your urine may look dark, thick, or cloudy. You may have fever, chills, nausea/vomiting, diarrhea, confusion, shortness of breath, irregular heartbeat, fatigue, muscle pain, joint discomfort, and/or seizure. If you notice any of these, tell your

doctor or nurse right away. Your study doctor will closely watch and treat you as needed to lower the risk of any serious changes in your blood or other complications of TLS. You may need to have extra blood tests or EKGs to check for signs of TLS.

You should wear ear plugs or other hearing protection when involved in a loud activity.

If you notice any rash, hives, itching, or other signs of an allergic reaction such as swelling, wheezing, or you are having a hard time breathing, tell your doctor right away.

Richter's Transformation (RT) is a change of chronic lymphocytic leukemia (CLL) into a more aggressive lymphoma. Richter's Transformation has happened to a small number of people that received venetoclax. It is not clear at this time if venetoclax treatment caused it to happen, or if it is a complication from your cancer.

## **Study Drug Combination Side Effects**

**Using the study drugs together** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

### Other Risks

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

Having **bone marrow aspirations/biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the aspiration/biopsy. An allergic reaction to the anesthetic may occur. A scar may form at the aspiration/biopsy site.

**X-rays** will expose you to radiation which can cause harm, such as burning or an increased risk of developing a cancer. Most radiation procedures use very small amounts of radiation. This is not expected to cause harm. These test amounts are not much different from exposures in usual daily life. However, the exposure risk is cumulative over a lifetime, and the total should be kept as low as possible.

**EKGs** may cause discomfort while lying on the exam table, and the tape on the EKG pads may cause skin irritation.

The type of **genetic testing** being performed in this study will not provide you or your doctor information about diseases that are passed down in families. It will not tell the study researchers anything that will prevent you from getting health insurance, and it will not tell the study researchers anything about any diseases or conditions you may get in the future.

This study may involve unpredictable risks to the participants.

# **Pregnancy Related Risks**

Because taking part in this study can result in risks to an unborn or breastfeeding baby, you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study and for at least 16 weeks after your last dose of study drug, if you are sexually active.

Birth Control Specifications: If you can become pregnant or father a child, you must use a double barrier method of birth control (2 forms of barrier birth control at the same time) and 1 other form of acceptable birth control while you are on this study and for at least 16 weeks after your last dose of study drug.

Acceptable methods of birth control are:

- Intrauterine devices (IUD) or intrauterine system (IUS), except IUD progesterone T
- Barrier method (such as a condom, diaphragm, or cervical/vault cap)
- Birth control pills, injections, or implants

Ask your doctor about acceptable forms of birth control.

Males: You should not donate sperm while you are on study and for at least 16 weeks after your last dose of study drug. Tell the doctor right away if your partner becomes pregnant or suspects pregnancy. Your partner will be asked to give consent to follow her pregnancy to the outcome.

Females: If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away.

Getting pregnant will result in your removal from this study.

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. There are no plans made by MD Anderson or Oncoceutics, Inc. to reimburse you for expenses or to compensate you financially for this injury.

If you suffer a study-related injury, you may contact the Chair of the study, Dr. Gautam Borthakur, at 713-563-1586, or 713-792-2121 (24-hours) with any questions you may have. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs, including hospitalization, nausea, vomiting, low blood cell

counts, and dehydration. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

# **Additional Information**

4. You may ask the study chair any questions you have about this study, if you have any questions, concerns, or complaints about the research, or if at any time you feel you have experienced a research-related injury or a reaction to the study drug. You may contact the study chair, Dr. Gautam Borthakur, at 713-563-1586, or 713-792-2121 (24-hours).

If you have questions about your rights as a research subject or if you have questions, concerns, or complaints about the research, you may contact:

WCG IRB

Telephone: 855-818-2289

E-mail: clientcare@wcgclinical.com

WCG IRB is a group of people who perform independent review of research.

WCG IRB will not be able to answer some study-specific questions, such as questions about appointment times. However, you may contact WCG IRB if the research staff cannot be reached or if you wish to talk to someone other than the research staff.

5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits to which you are otherwise entitled.

If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. If you withdraw from this study, you can still choose to be treated at MD Anderson.

- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, Oncoceutics, Inc., the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or WIRB.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.
- 9. This study is sponsored and/or supported by: Oncoceutics, Inc.
- 10. In a medical emergency, you may be cared for by someone who has a financial interest with the study sponsor(s). If you have any questions about this, you may call WIRB at 1-800-562-4789.
- 11. The MD Anderson Conflict of Interest policy states that MD Anderson employees may not serve as the study chair or co-chair on a research study if they have received funds that are greater than the amount allowed by the policy or own stock in the sponsoring or supporting companies.

The MD Anderson Conflict of Interest policy and the IRB require that you be told about significant financial relationships that the study staff and MD Anderson officials may have with the study sponsor(s).

At this time, no significant financial relationships with the study sponsor(s) have been disclosed by any of the study staff.

The following MD Anderson Conflicts of Interest exist:

MD Anderson and Oncoceutics, Inc. (the study sponsor) have an agreement for this study under which:

- Oncoceutics will provide the study drug for free for this study.
- If the study drug becomes commercially available, MD Anderson will receive part of the profit from the sale of this drug.
- If Oncoceutics is sold, MD Anderson will receive part of the money from the sale
- MD Anderson may also benefit financially if Oncoceutics chooses to buy out MD Anderson's rights to the study drug, ONC201, and its rights under its agreement with Oncoceutics.

You are being told about this relationship between MD Anderson and Oncoceutics because this is a conflict of interest.

MD Anderson has taken steps to help manage this conflict of interest. These steps are described in the Institutional Conflict of Interest Management and Monitoring Plan approved by the Executive Vice Chancellor for Health Affairs for The University of Texas System (EVC).

The plan requirements are listed below.

- Oversight of MD Anderson's two ONC201 clinical studies by an outside, independent Institutional Review Board (IRB)
- Review of safety and efficacy data by an outside, independent Data Safety Monitoring Board (DSMB)
- Periodic reporting to the EVC
- Disclosure of the MD Anderson financial interest to all clinical study patients, to all members of the ONC201 clinical studies research teams, and in all publications and oral presentations concerning the ONC201 clinical studies
- Posting of this summary on MD Anderson's public website
- Engagement of a non-MD Anderson ethicist to address any questions or Anderson financial interest and conflict of interest
- Referral of any concerns/complaints related to MD Anderson's compliance with the Institutional Conflict of Interest Management and Monitoring Plan, or its financial conflict of interest, to the Office of General Counsel for The University of Texas System
- Yearly review of MD Anderson's compliance with the Institutional Conflict of Interest Management and Monitoring Plan by The University of Texas System-wide Compliance Officer, with a written report of the review to be provided to the EVC

You will be given contact information for the outside, independent IRB.

MD Anderson will modify the Institutional Conflict of Interest Management and Monitoring Plan, if and when necessary, to address any future matters that may affect the integrity of the studies and to comply with any additional requirements thought necessary by the EVC to ensure the integrity of the studies.

This conflict of interest may affect your willingness to take part in this study. If you have any questions or concerns related to MD Anderson's financial relationship with Oncoceutics, please call the MD Anderson Institutional Compliance Office at 713-745-6636, and they will provide you with the contact information for a non-MD Anderson ethicist who can assist with your questions and concerns. In the event, a non-MD Anderson ethicist is not available, an MD Anderson ethicist will contact you to assist with your questions and concerns.

## **Future Research**

#### Data

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson and Oncoceutics, Inc., and/or shared with other researchers and/or institutions for use in future research.

### Samples

Samples (such as blood and/or tissue) are being collected from you as part of this study. Researchers at MD Anderson may use any leftover samples that are stored at MD Anderson in future research. Leftover samples stored by Oncoceutics, Inc. may be used in future research.

Before being used or shared for future research, every effort will be made to remove your identifying information from any data and/or research samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples.

#### **Genetic Research**

Research samples collected from you as part of this study may be used for genetic research, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment. If genetic research is done with your samples, those who have access to those samples may be able to identify you. The results of this research may also be able to be linked to you.

## **Authorization for Use and Disclosure of Protected Health Information:**

- **A.** During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Oncoceutics, Inc., and/or any future sponsors of the study
  - The EVC and the Office of General Counsel for The University of Texas System
  - Any future licensees of the study technology and an External Data Safety and Monitoring Board
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - WIRB
  - A non-MD Anderson ethicist
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it. If the results of this research are published, you will not be identified.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in in some situations, the FDA could be required to reveal the names of participants. If the results of this study are made public, information that identifies you will not be used.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI and it may be re-disclosed.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## **CONSENT/AUTHORIZATION**

I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I voluntarily agree to participate in this study. I authorize the release of my medical and research records for the purpose of this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed and dated copy of this consent document. SIGNATURE OF PARTICIPANT DATE PRINTED NAME OF PARTICIPANT PERSON OBTAINING CONSENT I have discussed this clinical research study with the participant, using language that is understandable and appropriate. I believe that I have fully informed this participant of the nature of this study and its possible benefits and risks and that the participant understood this explanation. PERSON OBTAINING CONSENT DATE

PRINTED NAME OF PERSON OBTAINING CONSENT